CLINICAL TRIAL: NCT03010683
Title: Effects of Agonists of Glucagon Like Peptide - 1 Receptors (GLP-1R) on Arterial Stiffness, Endothelial Glycocalyx and Coronary Flow Reserve in Patients With Coronary Artery Disease and Patients With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Associate Professor in Cardiology, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLP1-DM-ATTIKON
Record Dates: First submitted 2016-12-22; First posted 2017-01-05 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes Mellitus; Coronary Artery Disease
Keywords: Arterial stiffness; Endothelial glycocalyx; Coronary flow reserve
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Liraglutide; Metformin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- liraglutide (Active Comparator)
  Interventions: Drug: Liraglutide
- Metformin (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Liraglutide — Stimulation of Glucagon like peptide-1 receptor by liraglutide (Victoza) 1.8mg once daily as a subcutaneous injection
  Other Names: Victoza (liraglutide)
  Arms: liraglutide
Drug: Metformin — Antidiabetic drug-biguanide class (Glucophage) 1000mg twice daily per os
  Other Names: Glucophage (Metformin)
  Arms: Metformin

SUMMARY:
Arterial stiffness is associated with increased risk for cardiovascular disease. Moreover, the integrity of endothelial glycocalyx plays a vital role in vascular permeability, inflammation and elasticity. Agonists of Glucagon like peptide - 1 receptors (GLP-1R) used in the treatment of type 2 diabetes mellitus (T2DM). This category includes exenatide and liraglutide. These drugs lower glucose levels by inhibiting the secretion of glucagon, promoting the release of insulin in response to hyperglycemia, slowing gastric emptying, and augmenting satiety. Clinical studies have shown that GLP-1R agonists have beneficial effects on cardiovascular function in both diabetic patients and healthy subjects. The purpose of this study is to investigate in patients with T2DM without coronary artery disease (CAD), patients with T2DM and CAD and obese patients with abnormal oral glucose tolerance test (OGTT), changes in arterial stiffness, endothelial glycocalyx thickness and coronary reserve flow (CFR) after treatment with metformin or agonist GLP-1R.

DETAILED DESCRIPTION:
The investigators will study three groups matched for age and sex: 30 patients with type 2 diabetes mellitus (T2DM) without coronary artery disease (CAD), 30 patients with T2DM and CAD and 30 obese patients (BMI >30 Kg/m²) with abnormal oral glucose tolerance test (OGTT). It will be a randomized study with metformin or GLP-1R agonist treatment for 1 year. All subjects will receive for 1 year: (a) GLP-1R agonist or (b) metformin. At 0, 3, 6 and 12 months, where 0 is the starting point of treatment, blood samples will be collected.

At 0, 3, 6 and 12 months the investigators will measure:

1. Carotid-femoral pulse wave velocity (PWV, m/sec) using tonometry by Complior (SP ALAM) and augmentation index (AI, %) by the method of arteriography (Arteriograph, TensioMed)
2. Perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels (ranged from 5-25 micrometers) using Sideview Darkfield imaging (Microscan, Glycocheck). Increased PBR is considered an accurate non invasive index of reduced endothelial glucocalyx thickness.
3. Coronary flow reserve (CFR) in the left anterior descending artery after infusion of adenosine using Doppler echocardiography.
4. Determination of the following parameters in blood: glucose, insulin, free fatty acids, triglycerides, glycerol, C reactive protein (CRP), transforming growth factor-b (TGF-b), Lipoprotein-Associated Phospholipase A2 (LP-LPA2), tumor necrosis factor-a (TNF-a), interleukins 6 and 10 (IL6 and IL10), propeptide of type I procollagen (PIP), propeptide of procollagen type III (PIIINP), matrix metallopeptidases 9 and 2 (MMP), macrophage-colony stimulating factor (MCSF), growth differentiation factor-15 (GDF-15), N-terminal pro b-type natriuretic peptide (NT-proBNP) and galectin-3.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus (T2DM) without coronary artery disease (CAD)
* Patients with T2DM and CAD.
* Obese patients (BMI >30 Kg/m²) with abnormal oral glucose tolerance test (OGTT)

Exclusion Criteria:

* valvular heart disease
* congestive heart failure
* peripheral vascular disease
* liver or kidney failure
* history of alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; George Pavlidis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; Vaia Lambadiari, MD, Principal Investigator — 2nd Department of Internal Medicine, University of Athens, Greece; Fotini Kousathana, MD, Principal Investigator — 2nd Department of Internal Medicine, University of Athens, Greece; George Dimitriadis, MD, Principal Investigator — 2nd Department of Internal Medicine, University of Athens, Greece; John Lekakis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece
Locations (1):
- ''Attikon'' University General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595
- [Derived] Lambadiari V, Pavlidis G, Kousathana F, Varoudi M, Vlastos D, Maratou E, Georgiou D, Andreadou I, Parissis J, Triantafyllidi H, Lekakis J, Iliodromitis E, Dimitriadis G, Ikonomidis I. Effects of 6-month treatment with the glucagon like peptide-1 analogue liraglutide on arterial stiffness, left ventricular myocardial deformation and oxidative stress in subjects with newly diagnosed type 2 diabetes. Cardiovasc Diabetol. 2018 Jan 8;17(1):8. doi: 10.1186/s12933-017-0646-z. PMID 29310645

RESULTS

PARTICIPANT FLOW:
Groups:
- Liraglutide: Stimulation of glucagon like peptide-1 receptor by liraglutide (Victoza) 1.8 mg once daily as a subcutaneous injection
- Metformin: Antidiabetic drug - biguanide class (Glucophage) 1000 mg twice daily per os
Period: Overall Study
Arm/Group | Liraglutide | Metformin
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Metformin | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 6
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 7 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 20 | 20 | 40
Race/Ethnicity, Customized [Number; unit: participants]
  Greeks | 30 | 30 | 60
Pulse Wave Velocity [Mean (Standard Deviation); unit: m/s] | 11.8 (2.5) | 11.2 (3) | 11.5 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Differences in Pulse Wave Velocity at Baseline and 3, 6 and 12 Months After Treatment With Metformin or Agonist GLP-1R.
Description: Differences in carotid-femoral pulse wave velocity (PWV, m/sec) using tonometry at baseline and 3, 6 and 12 months after treatment with metformin or agonist GLP-1R.
Time Frame: Baseline, 3 months, 6 months and 12 months
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Liraglutide | Metformin
Number analyzed (Participants) | 30 | 30
m/s
  Baseline | 11.8 (2.5) | 11.2 (3)
  3 months | 11.6 (2.8) | 11.5 (2.7)
  6 months | 10.3 (3.3) | 11 (3)
  12 months | 10.5 (1.9) | 10.8 (2)

2. Primary Outcome: Differences in Augmentation Index at Baseline and 3, 6 and 12 Months After Treatment With Metformin or Agonist GLP-1R.
Description: Differences in augmentation index (AI, %) using oscillometry at baseline and 3, 6 and 12 months after treatment with metformin or agonist GLP-1R.
Time Frame: Baseline, 3 months, 6 months, and 12 months.
Measure: Mean (Inter-Quartile Range); unit: percentage of the central pulse pressure
Arm/Group | Liraglutide | Metformin
Number analyzed (Participants) | 30 | 30
percentage of the central pulse pressure
  Baseline | 18 [-1 to 31] | 14 [-9 to 24]
  3 months | 15.8 [-2 to 29] | 13.6 [-6 to 25]
  6 months | 13 [-2 to 31] | 15 [-8 to 24]
  12 months | 13.9 [-1 to 32] | 15.3 [-6 to 24]

3. Primary Outcome: Differences in Coronary Flow Reserve at Baseline and 3, 6 and 12 Months After Treatment With Metformin or Agonist GLP-1R.
Description: Differences in coronary flow reserve (CFR) using Doppler echocardiography at baseline and 3, 6 and 12 months after treatment with metformin or agonist GLP-1R.
Time Frame: Baseline, 3 months, 6 months, and 12 months.
Population: The investigators did not measure coronary flow reserve (CFR).
Arm/Group | Liraglutide | Metformin
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Differences in Endothelial Glycocalyx Thickness at Baseline and 3, 6 and 12 Months After Treatment With Metformin or Agonist GLP-1R.
Description: Differences in endothelial glycocalyx thickness as assessed by perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels at baseline and 3, 6 and 12 months after treatment with metformin or agonist GLP-1R. High PBR values represent reduced glycocalyx thickness.
Time Frame: Baseline, 3 months, 6 months, and 12 months.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Liraglutide | Metformin
Number analyzed (Participants) | 30 | 30
micrometers
  Baseline | 2.1 (0.29) | 2.13 (0.3)
  3 months | 2.07 (0.3) | 2.15 (0.3)
  6 months | 2.5 (0.2) | 2.13 (0.3)
  12 months | 2.04 (0.2) | 2.10 (0.3)

5. Secondary Outcome: Endothelial Glycocalyx and Pulse Wave Velocity.
Description: Association of endothelial glycocalyx thickness as assessed by perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels with pulse wave velocity (PWV, m/sec) at baseline and 3, 6 and 12 months after treatment with metformin or agonist GLP-1R.
Time Frame: Baseline, 3 months, 6 months, and 12 months.
Measure: Number; unit: Pearson correlation coefficient (r)
Arm/Group | Liraglutide | Metformin
Number analyzed (Participants) | 30 | 30
Pearson correlation coefficient (r)
  Baseline | 0.39 | 0.35
  3 months | 0.36 | 0.32
  6 months | 0.32 | 0.29
  12 months | 0.44 | 0.37

6. Secondary Outcome: Endothelial Glycocalyx and Coronary Flow Reserve.
Description: Association of endothelial glycocalyx thickness as assessed by perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels with coronary flow reserve (CFR) using Doppler echocardiography at baseline and 3, 6 and 12 months after treatment with metformin or agonist GLP-1R.
Time Frame: Baseline, 3 months, 6 months, and 12 months.
Population: The investigators did not estimate the association between endothelial glycocalyx thickness and coronary flow reserve (CFR) because they did not measure the CFR.
Arm/Group | Liraglutide | Metformin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Liraglutide | Metformin
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Οur study has a modest number of subjects. Additional large scale studies are needed to expand our results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT03010683/Prot_SAP_000.pdf